CLINICAL TRIAL: NCT03376178
Title: Ultrasound-guided Continuous Femoral Nerve Block: The Influence of Catheter Orifice Configuration (Six-hole Versus End-hole) on Post-operative Analgesia After Total Knee Arthroplasty. A Randomized Trial.
Brief Title: Catheter Orifice Configuration (Six-hole Versus End-hole) on Post-operative Analgesia After Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, FOURNIER ROXANE, MD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FROXANE
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Pain
Keywords: multiorifice or endhole femoral nerve catheter
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Eighty adult patients (aged ≥18 years) scheduled to undergo primary total knee arthroplasty under a combination of CFNB, sciatic nerve block and general anesthesia were randomized to CFNB using either a 3-pair micro-hole (Contiplex, BRAUN®, 20G - 400 mm) or an end-hole (Silverstim VYGON®, 20G - 500 mm) catheter. Once the femoral catheter was sited, a bolus of 20 mL lidocaine 1% was injected. An electronic pump then delivered an automated 5 mL bolus of ropivacaine 0.2% hourly, with 10 mL self-administered patient controlled analgesia boluses.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All investigators, patients, and other clinical staff were blinded to the treatment group. The investigator in charge of the patient was unaware of patient allocation. He did not perform the block or open the sealed and opaque envelope, but followed the patient in the ward. An opaque skin dressing was used in order to blind the type of catheter used. End-hole catheter Vygon is white and stiff whereas six-hole catheter contiplex is yellow and flexible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- six-hole group (Experimental): lidocaine and ropivacaine injection through catheters
  Interventions: Combination Product: lidocaine and ropivacaine injection through catheters
- end-hole group (Active Comparator): lidocaine and ropivacaine injection through catheters
  Interventions: Combination Product: lidocaine and ropivacaine injection through catheters

INTERVENTIONS:
Combination Product: lidocaine and ropivacaine injection through catheters — injection of local anesthetic through an endhole or a sixhole femoral nerve catheter in the context of total knee replacement. Analgesic properties at 24 and 48h of both groups registered.

SUMMARY:
Multiorifice catheters have been shown to provide superior analgesia and significantly reduce local anesthetic consumption compared with end-hole catheters in epidural studies. This prospective, blinded, randomized study tested the hypothesis that, in continuous femoral nerve block (CFNB) under ultrasound guidance, multiorifice catheter would reduce local anesthetic consumption at 24h compared with end-hole catheter.

DETAILED DESCRIPTION:
Eighty adult patients (aged ≥18 years) scheduled to undergo primary total knee arthroplasty under a combination of continuous femoral nerve block (CFNB), sciatic nerve block and general anesthesia were randomized to CFNB using either a 3-pair micro-hole (Contiplex, BRAUN®, 20G - 400 mm) or an end-hole (Silverstim VYGON®, 20G - 500 mm) catheter. Once the femoral catheter was sited, a bolus of 20 mL lidocaine 1% was injected. An electronic pump then delivered an automated 5 mL bolus of ropivacaine 0.2% hourly, with 10 mL self-administered patient controlled analgesia boluses.

ELIGIBILITY:
Inclusion Criteria:

* every patient accepting a conitnuous femoral nerve catheter

Exclusion Criteria:

* pregnancy,
* any contraindication to peripheral nerve blockade,
* pre-existing peripheral nerve neuropathy,
* allergy to LA (study medications),
* ASA score ≥4,
* neurologic or neuromuscular disease,
* psychiatric disease,
* renal failure,
* hepatic failure,
* chronic opioid therapy,
* NSAID contraindication,
* inability to use a patient controlled analgesia (PCA) device, g
* enu valgum,
* infection at the injection site or
* withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
total LA consumption at 24h | 24h after connecting PCA to the femoral nerve catheter
  total ropivacaine consumption at 24h in mL

SECONDARY OUTCOMES:
total LA consumption at 48h | 48h after connecting PCA to the femoral nerve catheter
  total ropivacaine consumption at 48h in mL
number of boluses of ropivacaine at 24h | 24h after connecting PCA to the femoral nerve catheter
  total ropivacaine boluses received at 24h in numbers
number of boluses of ropivacaine at 48 h | 48h after connecting PCA to the femoral nerve catheter
  total ropivacaine boluses received at 48h in numbers
quadriceps strength before surgery and 24h and 48h after surgery | quadriceps strenght before performing femoral nerve block and 24 and 48h after performing the block
  quadriceps strength measured with with an electronic dynamometer in N.m and percentage of preblock value of MVIC
morphine requirements at 24h and 48h | morphine consumption at 24h and 48h after completion of surgery
  rescue morphine 24h and 48h in mg

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tramer, Study Director — Anesthesiology department Of University Hospital of Geneva
Locations (1):
- University hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667
- [Background] Lang SA. Postoperative analgesia following total knee arthroplasty: a study comparing spinal anesthesia and combined sciatic femoral 3-in-1 block. Reg Anesth Pain Med. 1999 Jan-Feb;24(1):97. doi: 10.1016/s1098-7339(99)90176-1. No abstract available. PMID 9952105
- [Background] Farr J, Jaggers R, Lewis H, Plackis A, Sim SB, Sherman SL. Evidence-based approach of treatment options for postoperative knee pain. Phys Sportsmed. 2014 May;42(2):58-70. doi: 10.3810/psm.2014.05.2058. PMID 24875973
- [Background] Mizner RL, Snyder-Mackler L. Altered loading during walking and sit-to-stand is affected by quadriceps weakness after total knee arthroplasty. J Orthop Res. 2005 Sep;23(5):1083-90. doi: 10.1016/j.orthres.2005.01.021. Epub 2005 Mar 28. PMID 16140191
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Brodner G, Buerkle H, Van Aken H, Lambert R, Schweppe-Hartenauer ML, Wempe C, Gogarten W. Postoperative analgesia after knee surgery: a comparison of three different concentrations of ropivacaine for continuous femoral nerve blockade. Anesth Analg. 2007 Jul;105(1):256-62. doi: 10.1213/01.ane.0000265552.43299.2b. PMID 17578984
- [Background] Sia AT, Lim Y, Ocampo C. A comparison of a basal infusion with automated mandatory boluses in parturient-controlled epidural analgesia during labor. Anesth Analg. 2007 Mar;104(3):673-8. doi: 10.1213/01.ane.0000253236.89376.60. PMID 17312228
- [Background] Fredrickson MJ, Abeysekera A, Price DJ, Wong AC. Patient-initiated mandatory boluses for ambulatory continuous interscalene analgesia: an effective strategy for optimizing analgesia and minimizing side-effects. Br J Anaesth. 2011 Feb;106(2):239-45. doi: 10.1093/bja/aeq320. Epub 2010 Nov 25. PMID 21112881
- [Background] Fredrickson MJ, Ball CM, Dalgleish AJ. Catheter orifice configuration influences the effectiveness of continuous peripheral nerve blockade. Reg Anesth Pain Med. 2011 Sep-Oct;36(5):470-5. doi: 10.1097/AAP.0b013e318228d4ce. PMID 21857268
- [Background] Michael S, Richmond MN, Birks RJ. A comparison between open-end (single hole) and closed-end (three lateral holes) epidural catheters. Complications and quality of sensory blockade. Anaesthesia. 1989 Jul;44(7):578-80. doi: 10.1111/j.1365-2044.1989.tb11446.x. PMID 2774123
- [Derived] Novello-Siegenthaler A, Hamdani M, Iselin-Chaves I, Fournier R. Ultrasound-guided continuous femoral nerve block: a randomized trial on the influence of femoral nerve catheter orifice configuration (six-hole versus end-hole) on post-operative analgesia after total knee arthroplasty. BMC Anesthesiol. 2018 Dec 19;18(1):191. doi: 10.1186/s12871-018-0648-8. PMID 30567487